CLINICAL TRIAL: NCT07193212
Title: Osteopathic Manipulation Treatment Effect on the Leg and Foot Myofascial System in Adults With Chronic Low Back Pain - Pilot Study
Brief Title: How Osteopathic Treatment Affects the Leg and Foot in People With Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-206
Record Dates: First submitted 2025-09-08; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: chronic low back pain; myofascial systems; omt
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMT Treatment Group (Experimental)
  Interventions: Other: Osteopathic Manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Osteopathic Manipulative Treatment (OMT) is a hands-on approach where a trained physician uses techniques such as gentle pressure, stretching, and guided movements to improve mobility, reduce pain, and support the body's natural healing. It focuses on the interconnectedness of muscles, joints, and fascia to restore balance and function.

SUMMARY:
This pilot study will examine whether osteopathic manipulative treatment (OMT) can improve both physical and psychological aspects of chronic low back pain by focusing on the interconnected myofascial system of the back, legs, and feet. Twenty adults with chronic low back pain will receive four OMT sessions over 5-7 weeks. Before and after treatment, the investigators will measure muscle stiffness with ultrasound, plantar pressure during walking with a pressure plate, and patient-reported outcomes on pain, disability, sleep quality, stress, anxiety, depression, pain catastrophizing, and pain self-efficacy using surveys. By linking these objective and subjective measures, the study aims to provide early evidence of how OMT may influence musculoskeletal function, daily activity, and overall well-being, helping to guide future larger studies on treatment strategies for low back pain

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects 18-65 years old
* presence of chronic low back > 3 months duration or pain present > 50% of the time within the previous 12 months

Exclusion Criteria:

* prior surgery of the thoracic, lumbar or sacral spine, pelvis
* diagnosis lumbar radiculopathy or pinched nerve in the neck
* diagnosis of foot condition that alters gait
* diagnosis of connective tissue or muscle disorders
* diagnosis of cancer
* previous spinal cord injury inflammatory arthritis and fibromyalgia
* pregnancy
* tobacco use
* known diabetes or prediabetes
* allergy to ultrasound gel (propylene glycol)
* history of manual therapy treatment within the past 2 weeks
* injection for pain within the past 1 month
* currently taking muscle relaxers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stiffness of Low Back and Lower Extremity Muscles Assessed by Ultrasound Shear Wave Elastography | From baseline measures on Day 1 until the last OMT treatment, up to 6 weeks.
  Stiffness in the muscles of the low back and lower extremity will be quantitatively assessed using ultrasound shear wave elastography (SWE). SWE provides a non-invasive, reliable measure of tissue stiffness by calculating the shear wave speed (in meters/second) and corresponding elasticity modulus (in kilopascals). Regions of interest will be placed within target muscles and tissues (e.g., lumbar multifidus, thoracolumbar aponeurosis, hamstrings, gastrocnemius) and standardized acquisition protocols will be used to ensure reproducibility. This method allows for objective measurement of muscle stiffness rather than relying on subjective evaluation, thereby enhancing the validity of the outcome measure.
Body sway normalized path length, area, and velocity. | From baseline measures on Day 1 until the last OMT treatment, up to 6 weeks.
  A triaxial accelerometer will be used to measure postural control. The sensor will be secured over the lower trunk and measurements will occur under six conditions: feet together eyes open, feet together eyes closed, single-leg stance on the right and left with eyes opened and eyes closed. An average of 3 trials per condition will be used for each stance with 1 minute rest between trials. Double leg stance trials will be performed for 30 seconds while single leg stance trials will be performed for 15 seconds. Normalized path length (NPL) of acceleration in the anteroposterior (AP) and mediolateral (ML) directions, and sway excursion area, and velocity will be determined.

SECONDARY OUTCOMES:
Low back pain intensity and frequency. | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  Low back and lower extremity pain intensity, and frequency measured by an NRS (intensity) and Likert scale (frequency).
Functional disability. | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  The Roland-Morris Disability Questionnaire will be used to score functional disability.
Plantar Pressure Changes Assessed by EMED Pedobarographic Platform | From baseline measures on Day 1 until the last OMT treatment, up to 6 weeks.
  Plantar pressure distribution will be assessed using a validated EMED pedobarographic platform (Novel), which records dynamic foot pressures during gait. Outcome parameters will include peak pressure (kPa), pressure-time integrals, and center of pressure trajectory. Participants will walk barefoot at a self-selected pace across the platform, and standardized protocols will be used to ensure reproducibility. An average of 5 measures from each foot will be obtained.
Pain self-efficacy score | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  The pain self-efficacy questionnaire will be used to assess participants confidence in their ability to perform various activities and achieve goals despite experiencing pain, and its relationship to clinical response to treatment.

OTHER OUTCOMES:
Depression Assessed by Depression Anxiety Stress Scale-21 (DASS-21) | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  Depression will be assessed using the Depression Anxiety Stress Scale-21 (DASS-21), a validated 21-item self-report questionnaire. The Depression subscale consists of 7 items, each scored on a 4-point Likert scale (0 = did not apply to me at all; 3 = applied to me very much, or most of the time). Scores are summed and multiplied by two to yield a final subscale score ranging from 0 to 42, with higher scores reflecting greater depressive symptoms.
Anxiety Assessed by Depression Anxiety Stress Scale-21 (DASS-21) | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  Anxiety will be assessed using the DASS-21 questionnaire. The Anxiety subscale includes 7 items scored on a 4-point Likert scale (0-3). Subscale scores are summed and multiplied by two, yielding a final score from 0 to 42, with higher scores reflecting greater anxiety symptoms.
Stress Assessed by Depression Anxiety Stress Scale-21 (DASS-21) | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  Stress will be assessed using the DASS-21 questionnaire. The Stress subscale consists of 7 items scored on a 4-point Likert scale (0-3). Subscale scores are summed and multiplied by two, yielding a final score from 0 to 42, with higher scores reflecting greater stress symptoms.
Impact of sleep quality on daily function | From baseline measures on Day 1 until one week after the last OMT treatment, up to 7 weeks.
  The PROMIS Sleep-Related Impairment Short Form (8-item) will be used to assess changes in self-reported perceptions of daytime sleepiness, tiredness, and functional impairments related to poor sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cawley, DC, MS, MSHS, Principal Investigator — VCOM
Locations (1):
- Edward Via College of Osteopathic Medicine, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berenshteyn Y, Gibson K, Hackett GC, Trem AB, Wilhelm M. Is standing balance altered in individuals with chronic low back pain? A systematic review. Disabil Rehabil. 2019 Jun;41(13):1514-1523. doi: 10.1080/09638288.2018.1433240. Epub 2018 Jan 30. PMID 29382241
- [Background] Wang H, Zheng J, Fan Z, Luo Z, Wu Y, Cheng X, Yang J, Zhang S, Yu Q, Lo WLA, Wang C. Impaired static postural control correlates to the contraction ability of trunk muscle in young adults with chronic non-specific low back pain: A cross-sectional study. Gait Posture. 2022 Feb;92:44-50. doi: 10.1016/j.gaitpost.2021.11.021. Epub 2021 Nov 19. PMID 34823100
- [Background] Park J, Nguyen VQ, Ho RLM, Coombes SA. The effect of chronic low back pain on postural control during quiet standing: A meta-analysis. Sci Rep. 2023 May 16;13(1):7928. doi: 10.1038/s41598-023-34692-w. PMID 37193730
- [Background] Ruhe A, Fejer R, Walker B. Is there a relationship between pain intensity and postural sway in patients with non-specific low back pain? BMC Musculoskelet Disord. 2011 Jul 15;12:162. doi: 10.1186/1471-2474-12-162. PMID 21762484
- [Background] Ryum T, Stiles TC. Changes in pain catastrophizing, fear-avoidance beliefs, and pain self-efficacy mediate changes in pain intensity on disability in the treatment of chronic low back pain. Pain Rep. 2023 Sep 13;8(5):e1092. doi: 10.1097/PR9.0000000000001092. eCollection 2023 Sep. PMID 37719924
- [Background] Ogunlana MO, Odole AC, Adejumo A, Odunaiya N. Catastrophising, pain, and disability in patients with nonspecific low back pain. Hong Kong Physiother J. 2015 Dec;33(2):73-79. doi: 10.1016/j.hkpj.2015.03.001. Epub 2015 Apr 16. PMID 30930571
- [Background] Xu C, Fu Z, Wang J, Wu B, Wang XQ. Differences and Correlations of Anxiety, Sleep Quality, and Pressure-Pain Threshold between Patients with Chronic Low Back Pain and Asymptomatic People. Pain Res Manag. 2022 May 17;2022:8648584. doi: 10.1155/2022/8648584. eCollection 2022. PMID 35619991
- [Background] Nguyen C, Boutron I, Zegarra-Parodi R, Baron G, Alami S, Sanchez K, Daste C, Boisson M, Fabre L, Krief P, Krief G, Lefevre-Colau MM, Rannou F. Effect of Osteopathic Manipulative Treatment vs Sham Treatment on Activity Limitations in Patients With Nonspecific Subacute and Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2021 May 1;181(5):620-630. doi: 10.1001/jamainternmed.2021.0005. PMID 33720272
- [Background] Murillo C, Falla D, Rushton A, Sanderson A, Heneghan NR. Shear wave elastography investigation of multifidus stiffness in individuals with low back pain. J Electromyogr Kinesiol. 2019 Aug;47:19-24. doi: 10.1016/j.jelekin.2019.05.004. Epub 2019 May 3. PMID 31077992
- [Background] Menz HB, Dufour AB, Riskowski JL, Hillstrom HJ, Hannan MT. Foot posture, foot function and low back pain: the Framingham Foot Study. Rheumatology (Oxford). 2013 Dec;52(12):2275-82. doi: 10.1093/rheumatology/ket298. Epub 2013 Sep 17. PMID 24049103
- [Background] McClinton S, Weber CF, Heiderscheit B. Low back pain and disability in individuals with plantar heel pain. Foot (Edinb). 2018 Mar;34:18-22. doi: 10.1016/j.foot.2017.09.003. Epub 2017 Sep 28. PMID 29202429
- [Background] Loffler M, Schneider P, Schuh-Hofer S, Kamping S, Usai K, Treede RD, Nees F, Flor H. Stress-induced hyperalgesia instead of analgesia in patients with chronic musculoskeletal pain. Neurobiol Pain. 2022 Dec 6;13:100110. doi: 10.1016/j.ynpai.2022.100110. eCollection 2023 Jan-Jul. PMID 36561877
- [Background] Licciardone JC, Gatchel RJ, Aryal S. Recovery From Chronic Low Back Pain After Osteopathic Manipulative Treatment: A Randomized Controlled Trial. J Am Osteopath Assoc. 2016 Mar;116(3):144-55. doi: 10.7556/jaoa.2016.031. PMID 26927908
- [Background] Anukoolkarn K, Vongsirinavarat M, Bovonsunthonchai S, Vachalathiti R. Plantar Pressure Distribution Pattern during Mid-Stance Phase of the Gait in Patients with Chronic Non-Specific Low Back Pain. J Med Assoc Thai. 2015 Sep;98(9):896-901. PMID 26591401
- [Background] Alsaadi SM, McAuley JH, Hush JM, Maher CG. Prevalence of sleep disturbance in patients with low back pain. Eur Spine J. 2011 May;20(5):737-43. doi: 10.1007/s00586-010-1661-x. Epub 2010 Dec 29. PMID 21190045